CLINICAL TRIAL: NCT03576729
Title: Magnetic Resonance Spectroscopy (MRS) to Determine Neuroinflammation and Oxidative Stress in MPS I
Brief Title: MRS to Determine Neuroinflammation and Oxidative Stress in MPS I
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: Rare Diseases Clinical Research Network (Network); National Center for Advancing Translational Sciences (NCATS) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Lysosomal Disease Network (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00003680; U54NS065768 (NIH)
Record Dates: First submitted 2018-06-22; First posted 2018-07-03 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Mucopolysaccharidosis Type I
Keywords: Mucopolysaccharidosis type I; MPS I; MPS IH; MPS IHS; MPS IS; Mucopolysaccharidosis I
MeSH Terms: conditions — Mucopolysaccharidosis I

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hurler syndrome participants: Participants who have MPS IH, also called Hurler syndrome
- Hurler-Scheie/Scheie participants: Participants who have either MPS IHS or MPS IS. MPS IHS is also called Hurler-Scheie syndrome. MPS IS is also called Scheie syndrome.
- Healthy Controls: Age-matched healthy controls

SUMMARY:
Neuroinflammation and oxidative stress have been shown to be present in persons with mucopolysaccharidosis type I (MPS I), but their effect on disease severity and disease progression is unknown. The investigator intends to employ brain magnetic resonance spectroscopy (MRS), a non-invasive technique, along with analysis of neuroinflammation and oxidative stress biomarkers in the blood, to measure and determine the level of oxidative stress and neuroinflammation, and their impact on clinical variability in MPS I patients.

DETAILED DESCRIPTION:
Persons with MPS I have a wide range of clinical manifestations including central nervous system (CNS) impairment. The role of neuroinflammation and oxidative stress is one avenue of investigation which may clarify the broad neurological impairment in MPS I. Finding biomarkers that accurately describe the underlying and ongoing brain pathology is a key not only to understanding the disease, but also to understanding the possibility of new therapeutic approaches for MPS I patients.

The investigator will compare patients with Hurler syndrome, and Hurler-Scheie or Scheie syndrome, with healthy controls. There will be 10 participants in each group, resulting in a total of 30 participants. Within the Hurler-Scheie or Scheie syndrome group, the investigator will examine the association of clinical severity with the proposed measures. These findings might help determine whether hematopoietic cell transplantation (HCT), which is the treatment for Hurler syndrome patients, results in decreased oxidative stress and neuroinflammation as compared to Hurler-Scheie or Scheie syndrome patients, who are treated by enzyme replacement therapy (ERT). Additionally, these findings might help determine whether therapies directed at reducing neuroinflammation and oxidative stress in MPS I could enhance neurological outcomes.

Study hypothesis: neuroinflammation and oxidative stress are present in MPS I subjects and are reflective of disease severity.

ELIGIBILITY:
Inclusion Criteria:

MPS I participants must meet the following:

1. Diagnosis of Hurler syndrome, OR Hurler-Scheie syndrome, OR Scheie syndrome
2. 6 years of age or older at time of screening

Healthy control participants must meet all of the following:

1. Absence of neurological disorder
2. 6 years of age or older at time of screening

Exclusion Criteria:

Persons who have any of the following will not be enrolled in this study:

1. Any surgically implanted pacemaker
2. Any indwelling electronic device, including programmable shunts
3. Orthodontic braces, unless non-metallic
4. Other implanted metal in the body other than titanium
5. An inability or unwillingness to complete an MRI/MRS because of low cognitive function or behavioral dysregulation
6. Pregnancy

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 20 subjects who have MPS I and are 6 years of age or older will be recruited for this study: 10 with severe MPS I (post-HCT Hurler syndrome); and 10 with attenuated MPS I (Hurler Scheie or Scheie syndrome, and receiving ERT).
  In addition, 10 normal healthy controls, 6 years of age or older, will be recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Brain Magnetic Resonance Imaging/Magnetic Resonance Spectroscopy (MRI/MRS) | 1 day -Single encounter during an appointment which is set at time of study enrollment.
  In a single session, each participant will undergo unsedated brain magnetic resonance imaging/magnetic resonance spectroscopy (MRI/MRS) to determine the presence and extent of any brain neuroinflammation. These data will be acquired on the 7-Tesla Siemens Prisma scanner at the Center for Magnetic Resonance Research (CMRR) at the University of Minnesota in Minneapolis.

SECONDARY OUTCOMES:
Presence and Level of Neuroinflammatory Biomarker MIP-1alpha | 1 day -Single blood draw performed at the same time as the single neuroimaging encounter.
  The presence of macrophage inflammatory protein (MIP)-1α (MIP-1alpha) will be determined; and if present, the level of this inflammatory biomarker will be determined.
Presence and Level of Regulated and Normal T cell Expressed and Secreted (RANTES) | 1 day -Single blood draw performed at the same time as the single neuroimaging encounter.
  The presence of 'regulated and normal T cell expressed and secreted' (referred to as RANTES), alternatively also known as chemokine (C-C motif) ligand 5, or CCL5, will be determined. If present, the level of this inflammatory biomarker will be determined.
Presence and Level of Tumor Necrosis Factor Alpha (TNF-α) | 1 day -Single blood draw performed at the same time as the single neuroimaging encounter.
  The presence of tumor necrosis factor alpha (TNF-α) will be determined. If present, the level of this inflammatory biomarker will be determined.
Presence and Level of Interferon-gamma (IFN-γ) | 1 day -Single blood draw performed at the same time as the single neuroimaging encounter.
  The presence of interferon-gamma (IFN-γ) will be determined. If present, the level of this autoinflammatory biomarker will be determined.
Presence and Level of Interleukin 1 beta (IL1β) | 1 day -Single blood draw performed at the same time as the single neuroimaging encounter.
  The presence of interleukin 1 beta (IL1β) will be determined. If present, the level of this inflammatory biomarker will be determined.
Presence and Level of Interleukin 2 (IL2) | 1 day -Single blood draw performed at the same time as the single neuroimaging encounter.
  The presence of interleukin 2 (IL2) will be determined. If present, the level of this inflammatory biomarker will be determined.
Presence and Level of Interleukin 8 (IL8) | 1 day -Single blood draw performed at the same time as the single neuroimaging encounter.
  The presence of interleukin 8 (IL8), alternatively referred to as chemokine (C-X-C motif) ligand 8, or CXCL8, will be determined. If present, the level of this inflammatory biomarker will be determined.
Presence and Level of Total Glutathione | 1 day -Single blood draw performed at the same time as the single neuroimaging encounter.
  The presence of total glutathione will be determined. If present, the level of this antioxidant will be determined.
Determination of Blood Glutathione Redox Ratio | 1 day -Single blood draw performed at the same time as the single neuroimaging encounter.
  The blood glutathione redox ratio will be determined.
Presence and Level of Superoxide Dismutase (SOD) | 1 day -Single blood draw performed at the same time as the single neuroimaging encounter.
  The presence of superoxide dismutase (SOD) will be determined. If present, the level of this antioxidant will be determined.
Presence and Level of 8-isoprostane | 1 day -Single blood draw performed at the same time as the single neuroimaging encounter.
  The presence of 8-isoprostane will be determined. If present, the level of this inflammatory biomarker will be determined.
Presence and Levels of Thiobarbituric Acid Reactive Substances (TBARS) | 1 day -Single blood draw performed at the same time as the single neuroimaging encounter.
  The presence of thiobarbituric acid reactive substances (TBARS), which are biomarkers of the damage produced by oxidative stress, will be determined. If present, the levels of these biomarkers will be determined.
Presence and Level of 4-hydroxynonenal (4-HNE) | 1 day -Single blood draw performed at the same time as the single neuroimaging encounter.
  The presence of 4-hydroxynonenal (4-HNE) will be determined. If present, the level of this oxidative stress biomarker will be determined.
Presence and Level of Catalase | 1 day -Single blood draw performed at the same time as the single neuroimaging encounter.
  The presence of catalase will be determined. If present, the level of this oxidative stress biomarker will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Igor Nestrasil, PhD, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data is input to the NIH-funded Rare Diseases Clinical Research Network's Data Management & Coordinating Center ("DMCC"). Eventually this data will become part of the database of Genotypes and Phenotypes ("dbGaP"), which is part of the National Center for Biotechnology Information, U.S. National Library of Medicine.
Supporting Information: Study Protocol, CSR
Time Frame: De-identified individual data are input to the NIH-funded Rare Diseases Clinical Research Network's Data Management & Coordinating Center ("DMCC") as these data become available following participants' appointments. After the conclusion of this study and analysis of its data, these data will become part of the database of Genotypes and Phenotypes ("dbGaP"), which is part of the National Center for Biotechnology Information, U.S. National Library of Medicine. These data will remain available in this database indefinitely.
Access Criteria: Access criteria are determined by the National Center for Biotechnology Information, U.S. National Library of Medicine.

REFERENCES:
- [Background] Nestrasil I, Vedolin L. Quantitative neuroimaging in mucopolysaccharidoses clinical trials. Mol Genet Metab. 2017 Dec;122S:17-24. doi: 10.1016/j.ymgme.2017.09.006. Epub 2017 Sep 15. PMID 29111092
- [Background] Shapiro EG, Nestrasil I, Rudser K, Delaney K, Kovac V, Ahmed A, Yund B, Orchard PJ, Eisengart J, Niklason GR, Raiman J, Mamak E, Cowan MJ, Bailey-Olson M, Harmatz P, Shankar SP, Cagle S, Ali N, Steiner RD, Wozniak J, Lim KO, Whitley CB. Neurocognition across the spectrum of mucopolysaccharidosis type I: Age, severity, and treatment. Mol Genet Metab. 2015 Sep-Oct;116(1-2):61-8. doi: 10.1016/j.ymgme.2015.06.002. Epub 2015 Jun 17. PMID 26095521
- See also: Rare Diseases Clinical Research Network's web site — https://www.rarediseasesnetwork.org/LDN/